CLINICAL TRIAL: NCT00014209
Title: A Phase II Study Of Gemcitabine, Dexamethasone, And Cisplatin (GDP) In Patients With Either Hodgkin's Disease Or Aggressive Histology Non-Hodgkin's Lymphoma Which Is Relapsed Or Refractory
Brief Title: Combination Chemotherapy in Hodgkin's Disease or Non-Hodgkin's Lymphoma Not Responding to Previous Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY10; LILLY-CAN-NCIC-LY10 (Other: LILLY); CDR0000068518 (Other: PDQ)
Record Dates: First submitted 2001-04-10; First posted 2003-07-30 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Large-Cell, Anaplastic | interventions — Cisplatin; Dexamethasone; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: cisplatin
Drug: dexamethasone
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have Hodgkin's disease or non-Hodgkin's lymphoma that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of gemcitabine, dexamethasone, and cisplatin in patients with relapsed or refractory Hodgkin's disease or aggressive non-Hodgkin's lymphoma.
* Determine the qualitative and quantitative toxicity of this regimen in these two patient populations.

OUTLINE: This is a multicenter study. Patients are stratified according to disease (Hodgkin's disease vs non-Hodgkin's lymphoma).

Patients receive oral dexamethasone on days 1-4, cisplatin IV over 1 hour on day 1, and gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks, 3 months, and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 44-88 patients (22-44 per stratum) will be accrued for this study within 4-10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed Hodgkin's disease OR
* Histologically or cytologically confirmed aggressive non-Hodgkin's lymphoma (NHL) of B-cell origin (including immunoblastic, anaplastic large cell, mediastinal large B-cell, or T-cell rich B-cell NHL)

  * No prior diagnosis of low-grade NHL
  * No histologic evidence of transformation from indolent to aggressive histology
* Bidimensionally measurable disease that is clinically or radiologically documented

  * Bone lesions not considered bidimensionally measurable
  * Lymph nodes at least 1.5 cm by 1.5 cm OR
  * Other non-nodal lesions at least 1 cm by 1 cm
* Recurrent or refractory to 1 prior chemotherapy regimen (excluding gemcitabine and cisplatin)
* No known CNS involvement NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST or ALT no greater than 2.5 times ULN

Renal:

* Creatinine less than 1.6 mg/dL

Cardiovascular:

* No significant cardiac dysfunction or cardiovascular disease

Other:

* HIV negative
* No other concurrent or prior malignancy within the past 5 years except adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No other serious illness or medical condition that would preclude study
* No active uncontrolled bacterial, fungal, or viral infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior stem cell transplantation
* No concurrent monoclonal antibody therapy
* No concurrent growth factors during the first course of study

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior IV chemotherapy
* No prior cisplatin or gemcitabine
* No prior high-dose chemotherapy
* No other concurrent cytotoxic therapy

Endocrine therapy:

* No concurrent corticosteroids, except for physiologic replacement

Radiotherapy:

* No prior radiotherapy to more than 25% of functioning bone marrow
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* At least 2 weeks since prior major surgery

Other:

* No other concurrent anti-cancer therapy or experimental therapy

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2000-12-12 (Actual); Primary Completion 2002-07-15 (Actual); Study Completion 2009-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Crump, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada
Locations (13):
- Canada (13):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Moncton Hospital, Moncton, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Crump M, Baetz T, Couban S, Belch A, Marcellus D, Howson-Jan K, Imrie K, Myers R, Adams G, Ding K, Paul N, Shepherd L, Iglesias J, Meyer R. Gemcitabine, dexamethasone, and cisplatin in patients with recurrent or refractory aggressive histology B-cell non-Hodgkin lymphoma: a Phase II study by the National Cancer Institute of Canada Clinical Trials Group (NCIC-CTG). Cancer. 2004 Oct 15;101(8):1835-42. doi: 10.1002/cncr.20587. PMID 15386331
- [Result] Baetz T, Belch A, Couban S, Imrie K, Yau J, Myers R, Ding K, Paul N, Shepherd L, Iglesias J, Meyer R, Crump M. Gemcitabine, dexamethasone and cisplatin is an active and non-toxic chemotherapy regimen in relapsed or refractory Hodgkin's disease: a phase II study by the National Cancer Institute of Canada Clinical Trials Group. Ann Oncol. 2003 Dec;14(12):1762-7. doi: 10.1093/annonc/mdg496. PMID 14630682